CLINICAL TRIAL: NCT01355497
Title: Phase III, Randomized, Double-Blind, Placebo-Controlled Study of the Effect of GTx-024 on Muscle Wasting in Patients With Non-Small Cell Lung Cancer on First Line Platinum Plus a Non-Taxane Chemotherapy
Brief Title: Effect of GTx-024 on Muscle Wasting in Patients With Non-Small Cell Lung Cancer (NSCLC) on First Line Platinum
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G300505; POWER2 (Other: GTx)
Record Dates: First submitted 2011-05-12; First posted 2011-05-18 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Muscle Wasting; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Muscular Atrophy; Carcinoma, Non-Small-Cell Lung | interventions — ostarine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTx-024 3mg once daily (Experimental): subjects will be randomized to receive GTx-024 3mg sofgel capsule once daily for the duration of the trial
  Interventions: Drug: GTx-024
- placebo (Placebo Comparator): subjects will be randomized to receive matching placebo once daily for the duration of the trial
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GTx-024 — subjects will be randomized to receive GTx-024 3mg softgel for the duration of the trial.
  Other Names: enobosarm, ostarine
  Arms: GTx-024 3mg once daily
Drug: placebo — subject will receive matching placebo for the duration of the trial
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if the investigational drug GTx-024 can help patients with non small cell lung cancer increase physical function and maintain or gain muscle.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, multicenter, multinational efficacy and safety study in subjects with non small cell lung cancer. Subjects will be evenly randomized to placebo or GTx-024 prior to initiation of first line chemotherapy. The primary efficacy analysis will be based on total Lean Body Mass (LBM) and physical function.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary, signed informed consent in accordance with institutional policies
* be non-obese as defined as body mass index (BMI)< or = 32 and weight < 300 pounds (< 136 kg)
* have been diagnosed with Stage III or IV NSCLC
* be prior to first line chemotherapy
* planned first line chemotherapy regimen is platinum plus gemcitabine only or platinum plus vinorelbine only or platinum plus pemetrexed only
* if surgery is part of the cancer treatment, screening for this study should be conducted at least 4 weeks (28 days) after surgery
* life expectancy of > 6 months
* ECOG score < or = 1
* serum creatinine < or = 2.0 mg/dL
* MALES - age > or = 30 years
* - FEMALES - age >or=30 years and clinically confirmed as postmenopausal.Subjects must have undergone the onset of spontaneous or surgical menopause prior to the start of this study. Spontaneous menopause is defined as the natural cessation of ovarian function as indicated by being amenorrheic for at least 12 months. If the subject has been amenorrheic for >or=6 months but <12 months they must have a serum FSH concentration of >or=50 mIU/mL and an estradiol concentration of <or=25 pg/mL. Surgical menopause is defined as bilateral oophorectomy.
* MALES - subjects must agree to use a double barrier method of contraception during the study and for 3 months after study completion. This may include the following: condom + spermicide or condom + oral hormonal contraception
* MALES - have a serum PSA of < or = 4.0 ng/mL or a negative prostate biopsy (no prostate cancer) within 6 months of evaluation

Exclusion Criteria:

* Have, in the judgment of the Investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
* Have ALT/SGOT or AST/SGPT above 1.5 times the upper limit of normal (ULN) without evidence of liver metastases and above 5 times the ULN in subjects with evidence of liver metastases
* have alkaline phosphatase greater than 3 times ULN and/or total bilirubin levels above 2 mg/dL at baseline
* have biologic agents or kinase inhibitors as part of their first line chemotherapy regimen including, but not limited to bevacizumab (Avastin), gefitinib (Nexavar) and erlotinib (Tarceva)
* cardiovascular: uncontrolled hypertension, congestive heart failure or angina
* Pulmonary: Stage 4 chronic obstructive pulmonary disease (COPD)
* positive screen for Hepatitis B consisting of HBsAg (Hepatitis B Surface Antigen), unless subject was diagnosed > 10 years prior to enrollment and no evidence of active liver disease
* currently taking testosterone, oxandrolone (Oxandrin), testosterone-like agents (such as dehydroepiandrosterone (DHEA), androstenedione, and other androgenic compounds including herbals), or antiandrogens; previous therapy with testosterone and testosterone-like agents is acceptable with a 30 day washout (if previous testosterone therapy was long term depot within the past 6 months, the site should contact the medical monitor for this study to determine appropriate washout period)
* currently taking megestrol acetate (Megace), dronabinol (Marinol), medical marijuana (medical cannabis) or any prescription medication intended to increase appetite or treat unintentional weight loss
* have a baseline stair climb time >or=30 seconds (mean of two stair climbs)
* have active cancer, other than NSCLC or non-melanoma carcinoma of the skin, within the previous two years.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - GTx Investigative Site, Birmingham, Alabama
  - GTx Investigative Site, Scottsdale, Arizona
  - GTx Investigative Site, La Jolla, California
  - GTx Investigative Site, Long Beach, California
  - GTx Investigative Site, Miami, Florida
  - GTx Investigative Site, Orange City, Florida
  - GTx Investigative Site, Tampa, Florida
  - GTx Investigative Site, Decatur, Illinois
  - GTx Investigative Site, Peoria, Illinois
  - GTx Investigative Site, Skokie, Illinois
  - GTx Investigative Site, Goshen, Indiana
  - GTx Investigative Site, Indianapolis, Indiana
  - GTx Investigative Site, Ashland, Kentucky
  - GTx Investigative Site, Concord, Massachusetts
  - GTx Investigative Site, Saint Clair Shores, Michigan
  - GTx Investigative Site, Tupelo, Mississippi
  - GTx Investigative Site, Great Falls, Montana
  - GTx Investigative Site, Rochester, New York
  - GTx Investigative Site, Burlington, North Carolina
  - GTx Investigator, Flat Rock, North Carolina
  - GTx Investigative Site, Wilmington, North Carolina
  - GTx Investigative Site, Winston-Salem, North Carolina
  - GTx Investigative Site, Canfield, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - GTx Investigative Site, Sandusky, Ohio
  - GTx Investigative Site, Portland, Oregon
  - GTx Investigative Site, Lancaster, Pennsylvania
  - GTx Investigative Site, Spartanburg, South Carolina
  - GTx Investigative Site, Nashville, Tennessee
  - GTx Investigative Site, Round Rock, Texas

REFERENCES:
- [Derived] Crawford J, Prado CM, Johnston MA, Gralla RJ, Taylor RP, Hancock ML, Dalton JT. Study Design and Rationale for the Phase 3 Clinical Development Program of Enobosarm, a Selective Androgen Receptor Modulator, for the Prevention and Treatment of Muscle Wasting in Cancer Patients (POWER Trials). Curr Oncol Rep. 2016 Jun;18(6):37. doi: 10.1007/s11912-016-0522-0. PMID 27138015

RESULTS

PARTICIPANT FLOW:
Groups:
- GTx-024 3mg Once Daily: subjects will be randomized to receive GTx-024 for the duration of the trial
  GTx-024: subjects will be randomized to receive GTx-024 for the duration of the trial.
- Placebo: subjects will be randomized to matching placebo once daily for the duration of the trial
  placebo: subject will receive placebo for the duration of the trial
Period: Overall Study
Arm/Group | GTx-024 3mg Once Daily | Placebo
Started | 165 | 165
Completed | 99 | 102
Not Completed | 66 | 63
Not completed — Death | 19 | 18
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — other-not provided | 9 | 4
Not completed — Withdrawal by Subject | 12 | 20
Not completed — noncompliance | 1 | 2
Not completed — progressive disease | 11 | 8
Not completed — Adverse Event | 11 | 10

BASELINE CHARACTERISTICS:
Population: Subjects included in the Full Analysis Set
Groups:
- GTx-024: subjects will be randomized to receive GTx-024 for the duration of the trail
  GTx-024: subjects will be randomized to receive GTx-024 for the duration of the trial.
- Placebo: subjects will be randomized to receive placebo for the duration of the trial
  placebo: subject will receive placebo for the duration of the trial
- Total: Total of all reporting groups
Arm/Group | GTx-024 | Placebo | Total
Number analyzed (Participants) | 159 | 161 | 320
Age, Continuous [Median (Full Range); unit: years] | 60.0 [41 to 79] | 62.0 [40 to 81] | 61.0 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 114 | 113 | 227

OUTCOME MEASURES:

1. Primary Outcome: Physical Function
Description: Measure is the percentage of subjects at day 84 with stair climb power change >=10% from their baseline value.
Time Frame: Day 84
Population: Subjects included in the Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GTx-024 | Placebo
Number analyzed (Participants) | 159 | 161
percentage of subjects | 19.5 [13.6 to 26.5] | 24.8 [18.4 to 32.3]

2. Primary Outcome: Lean Body Mass
Description: Measure is the percentage of subjects at day 84 with lean body mass change >=0% from their baseline value.
Time Frame: Day 84
Population: Subjects included in the Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | GTx-024 | Placebo
Number analyzed (Participants) | 159 | 161
percentage of subjects | 46.5 [38.6 to 54.6] | 37.9 [30.4 to 45.9]

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: Initiation: 29 Nov 2011, Completion: 30 May 2013
Groups:
- Placebo Once Daily: subjects will be randomized to receive placebo for the duration of the trial
  placebo: subject will receive placebo for the duration of the trial
Arm/Group | GTx-024 3mg Once Daily | Placebo Once Daily
Serious Adverse Events (participants affected / at risk) | 109/165 | 113/165
Other Adverse Events (participants affected / at risk) | 149/165 | 157/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 3mg Once Daily (N=165) | Placebo Once Daily (N=165)
Anaemia (Blood and lymphatic system disorders) | 12 | 9
Neutropenia (Blood and lymphatic system disorders) | 10 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Hyperprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 1
Disease Progression (General disorders) | 18 | 26
Fatigue (General disorders) | 0 | 2
Sudden Death (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Condition Aggravated (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 5
Sepsis (Infections and infestations) | 1 | 2
Respiratory Tract Infection (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Infectious Pleural Effusion (Infections and infestations) | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Erosive Duodentitis (Gastrointestinal disorders) | 0 | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Mesentaric Artery Thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 6
Cognitive Disorder (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Neropathy Peripheral (Nervous system disorders) | 0 | 1
Optic Neuritis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Cardiac Failure (Cardiac disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 3
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Blood Urea Increased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 0 | 1
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1 (1)
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 3mg Once Daily (N=165) | Placebo Once Daily (N=165)
Anemia (Blood and lymphatic system disorders) | 84 (143) | 79 (119)
Neutropenia (Blood and lymphatic system disorders) | 51 (92) | 56 (114)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (45) | 29 (55)
Leukopenia (Blood and lymphatic system disorders) | 26 (39) | 28 (52)
Nausea (Gastrointestinal disorders) | 74 (153) | 73 (168)
Vomiting (Gastrointestinal disorders) | 45 (81) | 48 (82)
Constipation (Gastrointestinal disorders) | 21 (24) | 25 (33)
Diarrhoea (Gastrointestinal disorders) | 15 (25) | 17 (23)
Disease Progression (General disorders) | 29 (34) | 31 (36)
Fatigue (General disorders) | 26 (37) | 29 (41)
Asthenia (General disorders) | 25 (30) | 27 (35)
Pyrexia (General disorders) | 19 (25) | 20 (29)
Chest Pain (General disorders) | 6 (8) | 12 (14)
Oedema Peripheral (General disorders) | 7 (8) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 15 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 11 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (13)
Decreased Appetite (Metabolism and nutrition disorders) | 32 (38) | 28 (37)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 12 (15)
Blood Creatinine Increased (Investigations) | 23 (31) | 15 (22)
Dizziness (Nervous system disorders) | 14 (18) | 16 (18)
Headache (Nervous system disorders) | 14 (14) | 16 (20)
Pneumonia (Infections and infestations) | 10 (11) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (19) | 17 (19)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide Sponsor with an advance copy of any proposed results communication at least 60 days prior to the date of the planned submission or presentation and Sponsor shall have 60 days from receipt to request any changes. Sponsor may request a delay of up to 60 additional days.

The PI shall not present data until the earlier of Sponsor's publication of the results of all investigators participating in the Study or 18 months after completion of the Study at all participating sites.